CLINICAL TRIAL: NCT00085722
Title: The Efficacy of Prolotherapy in Osteoarthritic Knee Pain
Brief Title: Joint Injections for Osteoarthritic Knee Pain
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-2004-0112; K23AT001879-01 (NIH)
Record Dates: First submitted 2004-06-14; First posted 2004-06-16 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Osteoarthritis
Keywords: Injection Therapy
MeSH Terms: conditions — Osteoarthritis | interventions — Glucose; Sodium Chloride; Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dextrose (Experimental): Subjects in Group 1 receive PrT with 15% and 25% dextrose solution, as it is generally practiced in the US today.
  Interventions: Procedure: Dextrose Prolotherapy
- Normal saline (Placebo Comparator): Subjects in Group 2 will receive the same treatment as Group 1, except that a 0.9% 'normal' saline solution with no known benefit will be used instead of dextrose.
  Interventions: Procedure: Saline Prolotherapy
- Exercise (Other): At-home physical therapy exercises as a non-injection control
  Interventions: Other: At-home physical therapy exercise group

INTERVENTIONS:
Procedure: Dextrose Prolotherapy — Injection procedure: 50% dextrose is diluted with .9% 'normal' saline and 1% lidocaine to achieve 15% dextrose for ligament injections and 25% dextrose for intra-articular injection.
  Other Names: Dextrose
  Arms: Dextrose
Procedure: Saline Prolotherapy — 7 mL 9% 'normal' saline and 3mL 1% lidocaine
  Other Names: Saline
  Arms: Normal saline
Other: At-home physical therapy exercise group — Subjects in the at-home physical therapy exercise group will receive a patient information pamphlet about knee osteoarthritis and conservative care instructions for standard at-home physical therapy exercises
  Other Names: Exercise
  Arms: Exercise

SUMMARY:
The purpose of this study is to determine whether prolotherapy (PrT), a therapy based on injection of a sugar solution in and around the knee, can decrease pain and disability from knee osteoarthritis (OA).

DETAILED DESCRIPTION:
OA is a common, debilitating condition for which there is no cure and no known cause. Prolotherapy (PrT) is an injection-based therapy for chronic musculoskeletal pain in which an irritant solution is injected at painful ligaments and tendons to produce stronger connective tissue and decrease pain. Although limited studies suggest PrT is effective may be effective for low back pain, its use has not been rigorously studied in human clinical trials for osteoarthritis.

Participants in this study will be randomly assigned to receive one of three treatments: standard PrT, injections with a saline placebo, or a pamphlet with recommendations for home knee physical therapy. Injections will be given at Weeks 1, 5, and 9; injection group subjects will have the option to receive an additional 2 sets of injections. All participants will be assessed for a total of 1 year. A set of disease-specific and general quality-of-life questionnaires will be used to assess participants' outcomes . A randomized subset of participants (N=38)will receive magnetic resonance imaging (MRI)of the knee at baseline and 52 weeks. At study completion, participants who did not receive PrT will have the option to receive up to five sessions of PrT at no cost. Data will be collected for this group (minus MRI) and will be analyzed separately. Enrollment is limited to residents of Southern Wisconsin.

ELIGIBILITY:
Inclusion Criteria:

* Pain from knee osteoarthritis that has impacted life for 3 months to 10 years
* X-ray results indicating knee osteoarthritis

Exclusion Criteria:

* Knee osteoarthritis surgical candidate
* History of total knee joint repair
* Prior use of PrT
* Prior fracture of the knee joint
* Joint injection of steroids or other drugs within the past 3 months
* Rheumatoid or inflammatory arthritis
* Chronic use of narcotic medication
* Other chronic pain diagnoses
* diabetes mellitus
* Body mass index (BMI) greater than 45
* Unresolved litigation
* Pregnancy
* Co-morbidity that may interfere with the study

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2004-07; Primary Completion 2008-11-01 (Actual); Study Completion 2016-05-01 (Actual)

PRIMARY OUTCOMES:
Quality of life, pain scores and disability at wks 0, 5, 9, 12, 24, 52 | Participants will be followed for one year.

SECONDARY OUTCOMES:
Secondary outcomes include disease and general quality of life indicators (all subjects) and magnetic resonance image (in a subset of 37 subjects). | Participants will be monitored for one year.

CONTACTS AND LOCATIONS:
Overall Officials: David P. Rabago, MD, Principal Investigator — University of Wisconsin Dept of Family Medicine
Locations (2):
- United States (2):
  - Northeast Family Medical Center, Madison, Wisconsin
  - University of Wisconsin General Clinical Research Center, Madison, Wisconsin

REFERENCES:
- [Background] Rejeski WJ, Ettinger WH Jr, Shumaker S, Heuser MD, James P, Monu J, Burns R. The evaluation of pain in patients with knee osteoarthritis: the knee pain scale. J Rheumatol. 1995 Jun;22(6):1124-9. PMID 7674241
- [Background] Reeves KD, Hassanein K. Randomized, prospective, placebo-controlled double-blind study of dextrose prolotherapy for osteoarthritic thumb and finger (DIP, PIP, and trapeziometacarpal) joints: evidence of clinical efficacy. J Altern Complement Med. 2000 Aug;6(4):311-20. doi: 10.1089/10755530050120673. PMID 10976977
- [Background] Eberle E, Ottillinger B. Clinically relevant change and clinically relevant difference in knee osteoarthritis. Osteoarthritis Cartilage. 1999 Sep;7(5):502-3. doi: 10.1053/joca.1999.0246. No abstract available. PMID 10489324
- [Background] Klein RG, Eek BC, DeLong WB, Mooney V. A randomized double-blind trial of dextrose-glycerine-phenol injections for chronic, low back pain. J Spinal Disord. 1993 Feb;6(1):23-33. PMID 8439713
- [Background] Ongley MJ, Klein RG, Dorman TA, Eek BC, Hubert LJ. A new approach to the treatment of chronic low back pain. Lancet. 1987 Jul 18;2(8551):143-6. doi: 10.1016/s0140-6736(87)92340-3. PMID 2439856
- [Background] Dechow E, Davies RK, Carr AJ, Thompson PW. A randomized, double-blind, placebo-controlled trial of sclerosing injections in patients with chronic low back pain. Rheumatology (Oxford). 1999 Dec;38(12):1255-9. doi: 10.1093/rheumatology/38.12.1255. PMID 10587555
- [Background] Yelland MJ, Glasziou PP, Bogduk N, Schluter PJ, McKernon M. Prolotherapy injections, saline injections, and exercises for chronic low-back pain: a randomized trial. Spine (Phila Pa 1976). 2004 Jan 1;29(1):9-16; discussion 16. doi: 10.1097/01.BRS.0000105529.07222.5B. PMID 14699269
- [Background] Hackett GS, Hemwall GA, Montgomery GA. Ligament and Tendon Relaxation Treated by Prolotherapy. Fifth Ed. ed. Oak Park: Gustav A. Hemwall, 1993
- [Background] Linetsky FS, FRafael M,. Pain Management, 2002:381-402.
- [Background] Dorman TA. Prolotherapy: A survey. The Journal of Orthopaedic Medicine 1993;15(2):49-50
- [Background] Reeves KD, Hassanein K. Randomized prospective double-blind placebo-controlled study of dextrose prolotherapy for knee osteoarthritis with or without ACL laxity. Altern Ther Health Med. 2000 Mar;6(2):68-74, 77-80. PMID 10710805
- [Background] Rogers WH, Wittink H, Wagner A, Cynn D, Carr DB. Assessing individual outcomes during outpatient multidisciplinary chronic pain treatment by means of an augmented SF-36. Pain Med. 2000 Mar;1(1):44-54. doi: 10.1046/j.1526-4637.2000.99102.x. PMID 15101963
- [Derived] Rabago D, Patterson JJ, Mundt M, Zgierska A, Fortney L, Grettie J, Kijowski R. Dextrose and morrhuate sodium injections (prolotherapy) for knee osteoarthritis: a prospective open-label trial. J Altern Complement Med. 2014 May;20(5):383-91. doi: 10.1089/acm.2013.0225. Epub 2014 Mar 17. PMID 24635447
- [Derived] Rabago D, Patterson JJ, Mundt M, Kijowski R, Grettie J, Segal NA, Zgierska A. Dextrose prolotherapy for knee osteoarthritis: a randomized controlled trial. Ann Fam Med. 2013 May-Jun;11(3):229-37. doi: 10.1370/afm.1504. PMID 23690322
- [Derived] Rabago D, Zgierska A, Fortney L, Kijowski R, Mundt M, Ryan M, Grettie J, Patterson JJ. Hypertonic dextrose injections (prolotherapy) for knee osteoarthritis: results of a single-arm uncontrolled study with 1-year follow-up. J Altern Complement Med. 2012 Apr;18(4):408-14. doi: 10.1089/acm.2011.0030. PMID 22515800
- See also: University of Wisconsin Department of Family Medicine Web Site — http://www.fammed.wisc.edu/